CLINICAL TRIAL: NCT06844721
Title: Association Between Murray Law-Based Angiography-Derived Fractional Flow Reserve and Outcomes After Coronary Artery Bypass Grafting
Brief Title: Association Between ΜFR and CABG Outcomes
Status: Active, not recruiting | Type: Observational
Sponsor: Seoul National University Hospital (Other)
Collaborators: Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Ho Young Hwang, professor, Seoul National University Hospital
Other Study IDs: H-2212-151-1390
Record Dates: First submitted 2025-02-15; First posted 2025-02-25 (Actual); Last update posted 2025-02-25 (Actual); Status verified 2025-02

CONDITIONS: Coronary Artery Bypass Graft Surgery (CABG)
Keywords: quantitative flow reserve; coronary artery bypass graft surgery (CABG); graft patency; clinical outcomes

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The goal of this observational study is to evaluate the association between Murray law-based quantitative flow reserve and outcomes after coronary artery bypass graft surgery.

DETAILED DESCRIPTION:
The goal of this observational study is to evaluate the association between Murray law-based quantitative flow reserve and outcomes after coronary artery bypass graft surgery. By constructing registry database during 10-year periods, several types of study objectives including 'graft patency' and 'long-term clinical outcomes' will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

1. patients who underwent isolated off-pump CABG for 3-vessel disease,
2. patients who underwent preoperative coronary angiography that fits for μFR analysis,

Exclusion Criteria:

1. Patients who underwent on-pump CABG
2. Patients in whom quality of preoperative coronary angiography did not fit for μFR analysis

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 3VD patients who underwent isolated off-pump CABG
Sampling Method: Non-Probability Sample
Enrollment: 945 (Actual)
Dates: Start 2008-01-01 (Actual); Primary Completion 2025-03-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Graft patency rate | 1 year after surgery
  1 year graft patency rate after surgery
Number of participants with Long-term all-cause mortality | From date of enrollment (operation) until the date of death from any cause, assessed up to 15 years").
  All-cause mortality indicates death from any cause during follow-up

SECONDARY OUTCOMES:
Number of partipiciants with major adverse cardiac events | From date of enrollment (operation) until the date of first documented major events or date of death from any cause, whichever came first, assessed up to 15 years
  MACE includes death, repeat revascularization and non-fatal myocardial infraction

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Yes
There is a plan to make individual participant data (IPD) and related data dictionaries available.
Supporting Information: Study Protocol, SAP
Time Frame: Starting 6 months after publication
Access Criteria: IPD will be shared on reasonable request to the corresponding author.

REFERENCES:
- [Background] Kotoku N, Ninomiya K, Ding D, O'Leary N, Tobe A, Miyashita K, Masuda S, Kageyama S, Garg S, Leipsic JA, Mushtaq S, Andreini D, Tanaka K, de Mey J, Wijns W, Tu S, Piazza N, Onuma Y, Serruys PW. Murray law-based quantitative flow ratio to assess left main bifurcation stenosis: selecting the angiographic projection matters. Int J Cardiovasc Imaging. 2024 Jan;40(1):195-206. doi: 10.1007/s10554-023-02974-z. Epub 2023 Oct 23. PMID 37870715
- [Background] Tu S, Ding D, Chang Y, Li C, Wijns W, Xu B. Diagnostic accuracy of quantitative flow ratio for assessment of coronary stenosis significance from a single angiographic view: A novel method based on bifurcation fractal law. Catheter Cardiovasc Interv. 2021 May 1;97 Suppl 2:1040-1047. doi: 10.1002/ccd.29592. Epub 2021 Mar 4. PMID 33660921
- [Background] Tonino PA, De Bruyne B, Pijls NH, Siebert U, Ikeno F, van' t Veer M, Klauss V, Manoharan G, Engstrom T, Oldroyd KG, Ver Lee PN, MacCarthy PA, Fearon WF; FAME Study Investigators. Fractional flow reserve versus angiography for guiding percutaneous coronary intervention. N Engl J Med. 2009 Jan 15;360(3):213-24. doi: 10.1056/NEJMoa0807611. PMID 19144937
- [Background] Pijls NH, van Schaardenburgh P, Manoharan G, Boersma E, Bech JW, van't Veer M, Bar F, Hoorntje J, Koolen J, Wijns W, de Bruyne B. Percutaneous coronary intervention of functionally nonsignificant stenosis: 5-year follow-up of the DEFER Study. J Am Coll Cardiol. 2007 May 29;49(21):2105-11. doi: 10.1016/j.jacc.2007.01.087. Epub 2007 May 17. PMID 17531660
- [Derived] Hwang HY, Ding D, Kang J, Sun P, Sohn SH, Tu S, Koo BK. Association Between Angiography-Derived Murray Law-Based Quantitative Flow Ratio and 1-Year Coronary Artery Bypass Graft Patency. JACC Cardiovasc Interv. 2025 Oct 13;18(19):2326-2334. doi: 10.1016/j.jcin.2025.08.027. PMID 41093449